CLINICAL TRIAL: NCT06118515
Title: A Phase I Pharmacokinetic and Safety Assessment of Oral Letermovir in Infants With Symptomatic Congenital Cytomegalovirus Disease
Brief Title: A Safety Assessment of Oral Letermovir in Infants With Symptomatic Congenital Cytomegalovirus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-0027; 5U54AI150225-05 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07-18

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Congenital Cytomegalovirus Disease; Infants; Letermovir; Pharmacokinetic; Phase 1
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Neonates (</= 83 days) with symptomatic congenital Cytomegalovirus (CMV) disease will receive one dose of oral letermovir, using weight dose banding. All subjects also will receive valganciclovir as standard of care. A dose safety evaluation will occur to ensure the safety data support subjects proceeding. If the observed letermovir exposure is </= 100,000 ngxhr/mL, the subject will initiate a 14-day course of once-daily oral letermovir at the same dose as utilized on the Dose Finding Day. If the observed letermovir exposure of the subject is > 100,000 ngxhr/mL, the once-daily oral letermovir dose that will be used will be adjusted down in 2.5 mg increments from the dose utilized on the Dose Finding Day. N = 4
  Interventions: Drug: Letermovir
- Group 2 (Experimental): Neonates (</= 90 days) with symptomatic congenital Cytomegalovirus (CMV) disease will initiate a 14-day course of once-daily oral letermovir, using weight dose banding. All subjects also will receive valganciclovir as standard of care. A dose escalation safety evaluation will occur to ensure the safety data support subjects proceeding. If the median of observed letermovir exposures of subjects in Group 1 is below 34,400 ngxhr/mL (or above 100,000 ngxhr/mL), then the subjects enrolled in Group 2 will receive once-daily oral letermovir at a dose that has been adjusted upward (or downward) in 2.5 mg increments. N=8
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Letermovir is a novel inhibitor targeting the cytomegalovirus (CMV) viral enzyme, effectively disrupting the production of additional CMV virions. Letermovir has demonstrated potent, selective, and reversible inhibition of CMV activity in preclinical studies.

SUMMARY:
This is a Phase 1 single-arm open-label study of letermovir in neonates with symptomatic congenital Cytomegalovirus (CMV) disease. There will be two groups enrolled. Group 1 will be comprised of 4 subjects. Following documentation study inclusion and signing of informed consent, Group 1 subjects will receive one dose of oral letermovir (Study Day 0), using the dose bands. A full pharmacokinetics (PK) profile will then be obtained over the next 24 hours, and blood specimens will be shipped immediately to the University of Alabama at Birmingham (UAB) Pharmacokinetic Lab and processed in real time. Within = 7 days, pharmacokinetics (PK) results will be conveyed to the study site. If the Area Under the Curve (AUC24) is =100,000 ngxhr/mL (see footnote a in Table 1), the subject will initiate a 14-day course of once-daily oral letermovir at the same dose as utilized on Dose Finding Day. This duration of letermovir therapy was selected based upon our earlier observation in this population that patients with symptomatic congenital Cytomegalovirus (CMV) disease who achieve viral suppression to =2.5 log by day 14 of valganciclovir therapy and then maintain it over the next 4 months are statistically more likely to have improved hearing across the first two years of life (22). If the observed letermovir exposure of the subject is > 100,000 ngxhr/mL, the once-daily oral letermovir dose that will be used will be adjusted down in 2.5 mg increments. Oral valganciclovir (16 mg/kg/dose BID) will begin within the first month of life, as standard of care; initiation of valganciclovir can be concomitant with or prior to initiation of the 14-day course of letermovir (but will not start before obtaining the pharmacokinetics (PK) specimens following the single dose of letermovir on the Dose Finding Day). This is similar to the intensification approach that has been evaluated in the management of patients infected with human immunodeficiency virus (23-25). The day that the 14-day course of letermovir begins for Group 1 subjects will be known as Study Day 1. Serial blood samples will be obtained on Study Days 1, 5, 10, and 14 for safety chemistry and hematology labs and for Cytomegalovirus (CMV) viral loads. Cytomegalovirus (CMV) viral load will be followed as well on Study Days 21 and 42 to assess for rebound in Cytomegalovirus (CMV) following cessation of letermovir treatment on Study Day 14. Saliva and urine viral loads will be followed at these timepoint as well. Full pharmacokinetics (PK) profiles for both letermovir and ganciclovir will be obtained on Study Day 10. In addition, sparse pharmacokinetics (PK) sampling will be obtained on Study Days 1, 5, and 14. Adverse events will be assessed at each study visit during treatment, and at Study Days 21 and 42 (4 weeks after the last study drug dose). Subjects then will continue on oral valganciclovir as routine clinical care to complete an anticipated 6 month duration of total therapy. The primary Objective is to determine the systemic exposure (AUC24) of letermovir following administration of oral letermovir granules in infants with symptomatic congenital CMV disease.

DETAILED DESCRIPTION:
This is a Phase 1 single-arm open-label study of letermovir in neonates with symptomatic congenital Cytomegalovirus (CMV) disease. There will be two groups enrolled. Group 1 will be comprised of 4 subjects. Following documentation study inclusion and signing of informed consent, Group 1 subjects will receive one dose of oral letermovir (Study Day 0), using the dose bands. A full pharmacokinetics (PK) profile will then be obtained over the next 24 hours, and blood specimens will be shipped immediately to the University of Alabama at Birmingham (UAB) Pharmacokinetic Lab and processed in real time. Within = 7 days, pharmacokinetics (PK) results will be conveyed to the study site. If the Area Under the Curve (AUC24) is =100,000 ngxhr/mL (see footnote a in Table 1), the subject will initiate a 14-day course of once-daily oral letermovir at the same dose as utilized on the Dose Finding Day. This duration of letermovir therapy was selected based upon our earlier observation in this population that patients with symptomatic congenital Cytomegalovirus (CMV) disease who achieve viral suppression to =2.5 log by day 14 of valganciclovir therapy and then maintain it over the next 4 months are statistically more likely to have improved hearing across the first two years of life (22). If the observed letermovir exposure of the subject is > 100,000 ngxhr/mL, the once-daily oral letermovir dose that will be used will be adjusted down in 2.5 mg increments. Oral valganciclovir (16 mg/kg/dose BID) will begin within the first month of life, as standard of care; initiation of valganciclovir can be concomitant with or prior to initiation of the 14-day course of letermovir (but will not start before obtaining the pharmacokinetics (PK) specimens following the single dose of letermovir on the Dose Finding Day). This is similar to the intensification approach that has been evaluated in the management of patients infected with human immunodeficiency virus (23-25). The day that the 14-day course of letermovir begins for Group 1 subjects will be known as Study Day 1. Serial blood samples will be obtained on Study Days 1, 5, 10, and 14 for safety chemistry and hematology labs and for Cytomegalovirus (CMV) viral loads. Cytomegalovirus (CMV) viral load will be followed as well on Study Days 21 and 42 to assess for rebound in Cytomegalovirus (CMV) following cessation of letermovir treatment on Study Day 14. Saliva and urine viral loads will be followed at these timepoint as well. Full pharmacokinetics (PK) profiles for both letermovir and ganciclovir will be obtained on Study Day 10. In addition, sparse pharmacokinetics (PK) sampling will be obtained on Study Days 1, 5, and 14. Adverse events will be assessed at each study visit during treatment, and at Study Days 21 and 42 (4 weeks after the last study drug dose). Subjects then will continue on oral valganciclovir as routine clinical care to complete an anticipated 6 month duration of total therapy. Following enrollment of the 4 subjects in Group 1, the Safety Monitoring Committee (SMC) will review all safety and pharmacokinetic data. If no halting rules are met and no other safety concerns are identified, then additional subjects will be enrolled in Group 2. Subjects in Group 2 will initiate a 14-day course of once-daily oral letermovir, using the dose bands listed in Table 1, at the same time that oral valganciclovir (16 mg/kg/dose BID) is initiated as standard of care; initiation of valganciclovir can be concomitant with or prior to initiation of the 14-day course of letermovir. If the median of observed letermovir exposures of subjects in Group 1 is below 34,400 ngxhr/mL (or above 100,000 ngxhr/mL), then the subjects enrolled in Group 2 will receive once-daily oral letermovir at a dose that has been adjusted upward (or downward) in 2.5 mg increments. The day that the 14-day course of letermovir begins for Group 2 will be known as Study Day 1. Serial blood samples will be obtained on Study Days 1, 5, 10, and 14 for safety chemistry and hematology labs and for Cytomegalovirus (CMV) viral loads. Cytomegalovirus (CMV) viral load will be followed as well on Study Days 21 and 42 to assess for rebound in Cytomegalovirus (CMV) following cessation of letermovir treatment on Study Day 14. Saliva and urine viral loads will be followed at these timepoint as well. Full pharmacokinetics (PK) profiles for both letermovir and ganciclovir will be obtained on Study Day 10. In addition, sparse pharmacokinetics (PK) sampling will be obtained on Study Days 1, 5, and 14. Adverse events will be assessed at each study visit during treatment, and at Study Days 21 and 42 (4 weeks after the last study drug dose). Subjects then will continue on oral valganciclovir as routine clinical care to complete an anticipated 6 month duration of total therapy. The primary Objective is to determine the systemic exposure (AUC24) of letermovir following administration of oral letermovir granules in infants with symptomatic congenital CMV disease. the secondary objectives are 1.) To determine the other pharmacokinetic parameters of letermovir following administration of oral letermovir granules in infants with symptomatic congenital CMV disease; 2.) To evaluate the safety of letermovir oral granules in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent(s) or legal guardian(s)
2. Cytomegalovirus (CMV) confirmation by culture, shell vial, or Polymerase Chain Reaction (PCR) tests from a specimen obtained at </= 30 days of life from saliva, blood, or urine
3. Symptomatic congenital CMV disease*
4. Age at study enrollment:

   1. </= 83 days for Group 1 subjects**
   2. </= 90 days for Group 2 subjects
5. Weight at study enrollment 2.6 kg to < 8.0 kg
6. Gestational age >/= 32 weeks at birth
7. Intention by patient's physician to clinically treat infant with oral valganciclovir for 6 months for symptomatic congenital CMV disease

   * Manifested by one or more of the following: thrombocytopenia; petechiae; hepatomegaly; splenomegaly; intrauterine growth restriction; hepatitis; or Central Nervous System (CNS) involvement such as microcephaly, radiographic abnormalities indicative of CMV CNS disease, abnormal cerebrospinal fluid (CSF) indices for age, chorioretinitis, hearing deficits as detected by formal brainstem evoked response, and/or positive CMV Polymerase Chain Reaction (PCR) from CSF **Group 1 subjects must enroll and receive the Dose Finding Day dose of letermovir on or before 83 days of life so that oral valganciclovir can be started prior to 12 weeks 6 days (which is 90 days) of life, as is standard of care. For this study, the date of birth is counted as day of life 0

Exclusion Criteria:

1. Imminent demise
2. Infants known to be born to women who are HIV positive (but HIV testing is not required for study entry)
3. Current receipt of other investigational drugs
4. Grade 3 or 4 alanine aminotransferase (ALT) utilizing Division of AIDS (DAIDS) Toxicity Table
5. Grade 3 or 4 total bilirubin utilizing DAIDS Toxicity Table
6. Gastrointestinal abnormality which might preclude absorption of an oral medication (e.g., a history of necrotizing enterocolitis)
7. Anticipated concomitant administration of carbamazepine (Tegretol), nafcillin, phenobarbital, or phenytoin (Dilantin) during the period of study drug administration

Ages: 0 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Plasma letermovir area under the curve (AUC24) concentrations | Through Day 14
  Determined using the linear-log trapezoidal rule. In addition, a population PK analysis may be conducted at the end of the study.

SECONDARY OUTCOMES:
Frequency of serious adverse events (SAEs) | Through Day 14
Frequency of grade 3 adverse events (AEs) | Through Day 14
  Grade 3 is defined as severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated
Frequency of grade 4 adverse events (AEs) | Through Day 14
  Grade 4 is defined as Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death
Plasma letermovir clearance (CL) | Through Day 14
Plasma letermovir half-life (T1/2) | Through Day 14
  Determined using regression analysis of the terminal elimination phase concentration-time points.
Plasma letermovir maximum plasma concentration (Cmax) | Through Day 14
Plasma letermovir minimum plasma concentration (Cmin) | Through Day 14
Plasma letermovir volume of distribution (Vd) | Through Day 14

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Children's of Alabama Child Health Research Unit (CHRU), Birmingham, Alabama
  - Children's National Medical Center - Sheikh Zayed Campus - Infectious Disease, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Louisville School of Medicine - Norton Children's Hospital - Infectious Diseases, Louisville, Kentucky
  - Louisiana State University Health Shreveport - Infectious Diseases, Shreveport, Louisiana
  - University of Minnesota - Pediatric Infectious Disease, Minneapolis, Minnesota
  - SUNY Upstate Medical University Hospital - Pediatrics, Syracuse, New York
  - Nationwide Children's Hosp.-Neonatology-Ctr. for Perinatal Rsrch., Columbus, Ohio
  - University of Texas Southwestern Medical Center - Pediatrics, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

DOCUMENTS (2):
  • Informed Consent Form: Group 1 (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT06118515/ICF_000.pdf
  • Informed Consent Form: Group 2 (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT06118515/ICF_001.pdf